CLINICAL TRIAL: NCT06529718
Title: A Randomised, Phase II Trial to Evaluate the Efficacy of Ivonescimab, a PD 1/VEGF Bispecific Antibody, Versus FOLFOX as Second Line Therapy for Locally Advanced/Metastatic Biliary Cancers
Brief Title: Testing Ivonescimab Versus FOLFOX in Advanced Biliary Tract Cancer Patients
Acronym: SEVILLA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Cancer Research UK & UCL Cancer Trials Centre (Other); Belgian Group of Digestive Oncology (Other); Summit Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-GIG-2404 - PRODIGE 110; 2024-515875-36-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Biliary Tract Cancer
Keywords: Biliary tract cancer; Gallbladder; Cholangiocarcinoma
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma | interventions — Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Experimental treatment under study
  Interventions: Drug: Ivonescimab
- Control (Active Comparator): Standard of care second-line treatment for advanced biliary tract cancer
  Interventions: Drug: FOLFOX regimen

INTERVENTIONS:
Drug: Ivonescimab — 20 mg/kg IV infusion every 3 weeks
  Arms: Experimental
Drug: FOLFOX regimen — oxaliplatin 85 mg/m² IV, leucovorin 200 mg/m² IV (or folinic acid 400 mg/m²), and fluorouracil (5-FU) 400 mg/m² IV bolus; followed by 5 FU 2400 mg/m² as a 46 hour continuous IV infusion, every 2 weeks
  Arms: Control

SUMMARY:
The object of this trial is to test whether ivonescimab is superior to standard chemotherapy (FOLFOX regimen) for the treatment of patients with advanced biliary tract cancer after failure of a first line of chemotherapy. It is only open to patients who participated in the SAFIR-ABC10 trial (NCT05615818) but did not receive experimental treatment.

Eligible patients will be randomised (2:1) to receive either ivonescimab or FOLFOX. Treatment will be continued until disease progression, or a maximum of 34 cycles of ivonescimab (experimental arm), whichever occurs first.

DETAILED DESCRIPTION:
This is a Phase 2, multicentre, randomised, two-arm, open-label trial to evaluate whether ivonescimab is superior to standard second-line chemotherapy in the treatment of patients with advanced biliary tract cancer.

The trial will be open to patients who participated in the screening phase of the SAFIR-ABC10 protocol (NCT05615818) and who experienced disease progression on or following the first-line standard of care (CISGEM regimen).

A total of 72 patients will be enrolled and randomly assigned (2:1) to receive treatment with either:

* Experimental arm: Ivonescimab 20 mg/kg by intravenous infusion (IV) once every 3 weeks (Q3W).
* Control arm: Standard second-line chemotherapy - FOLFOX regimen Response to treatment will be assessed according to RECIST v1.1 by radiographic exams performed every 42 (±7) days. Patients will continue treatment until disease progression or for a maximum of 34 cycles of ivonescimab (experimental arm), whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Signed a written informed consent form prior to any trial specific procedures.
2. Histologically-proven intrahepatic cholangiocarcinoma, perihilar / distal cholangiocarcinoma, or gallbladder carcinoma (ampullary carcinoma excluded).
3. Locally advanced (non-resectable) or metastatic disease.
4. Participated in the Screening phase of the SAFIR-ABC10 trial.
5. Progression after first line standard of care (1L-SoC) regimen (CISGEM ± immunotherapy) as assessed by the investigator.
6. Eligible for second-line treatment with FOLFOX.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Presence of at least one evaluable lesion according to RECIST v1.1.
9. Age ≥18 years.
10. Adequate bone marrow function: absolute neutrophil count (ANC) ≥2 × 10⁹/L, platelet count ≥100 × 10⁹/L, and haemoglobin ≥9 g/dL.

    Note: Blood transfusion or growth factor therapy should not be performed within 7 days prior to the screening haematology analysis.
11. Adequate liver function: total bilirubin level ≤1.5 × the upper limit of normal (ULN) range (≤3 x ULN for patients with liver metastases or confirmed/suspected Gilbert syndrome, and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤2.5 × ULN (AST and ALT ≤5 x ULN when documented liver metastasis).
12. Adequate renal function: estimated creatinine clearance ≥50 mL/min according to the Cockcroft-Gault formula, or estimated glomerular filtration rate value ≥50 mL/min using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation, and urine protein < 2+ or 24 hour urine protein quantification < 1.0 g.
13. Coagulation: prothrombin time (PT) or international normalized ratio (INR) ≤ 1.5 x ULN, and partial prothrombin time (PTT) or activated PTT ≤ 1.5 × ULN (unless abnormalities are unrelated to coagulopathy,or prophylactic coagulation).
14. Adequate cardiac function: left ventricular ejection fraction (LVEF) ≥50% at baseline as determined by either echocardiogram or multigated acquisition (MUGA) scan.
15. Documented virology status of hepatitis, as confirmed by screening hepatitis B virus (HBV) and hepatitis C virus (HCV) tests: For patients with active HBV: HBV DNA <500 IU/ml during screening, initiation of anti-HBV treatment at least 14 days prior to randomization and willingness to continue anti-HBV treatment during the study (per local standard of care; e.g., entecavir). For patients with HCV, either with resolved infection (as evidenced by detectable antibody) or chronic infection (as evidence by detectable HCV RNA), are eligible.
16. Performance of an esophagogastroduodenoscopy within 6 months of inclusion and assessment and treatment of varices of all sizes per local standard of care prior to randomisation.
17. Biliary tract obstruction has been relieved.
18. Adequate biliary drainage, with no evidence of ongoing infection.
19. Women of childbearing potential (WOCBP) having sex with an unsterilized male partner and unsterilized males having sex with a female partner of childbearing potential, must agree to use an effective method of contraception for the duration of trial participation and as required after completing study treatment. Men must also agree to not donate sperm and women must agree to not donate oocytes during the specified period.
20. WOCBP must have a negative serum pregnancy test performed within 3 days before randomisation and a negative urine pregnancy test on the day of first dose, prior to treatment administration.
21. Willing and able to comply with the protocol for the duration of the study including scheduled visits, treatment plan, laboratory tests, and other study procedures.
22. Affiliated to a social security system or in possession of equivalent private health insurance (according to local regulations for participation in clinical trials).

Exclusion Criteria:

1. Toxicities from 1L-SoC not resolved to Grade ≤ 1 (according to version 5.0 of the National Cancer Institute - Common terminology criteria for adverse events [NCI-CTCAE v5.0]) before randomisation with the exception of alopecia.
2. Received first-line maintenance therapy with a matched target therapy proposed in SAFIR ABC10, or any second-line treatment.
3. Contraindication to ivonescimab.
4. Proven complete deficiency of dihydropyrimidine dehydrogenase (DPD).
5. Treatment with brivudine, sorivudine or their chemical analogues in the 4 weeks prior to randomisation.
6. Major surgical procedures or serious trauma within 4 weeks prior to randomisation, or plans for major surgery within 4 weeks after the first dose (as determined by the investigator). Minor local procedures (excluding central venous catheterisation and port implantation) within 3 days prior to randomisation.
7. History of bleeding tendencies or coagulopathy and/or clinically significant bleeding symptoms or risk within 4 weeks prior to randomisation, including but not limited to:

   1. Gastrointestinal bleeding.
   2. Haemoptysis (defined as coughing up ≥ 0.5 teaspoon of fresh blood or small blood clots).

      Note: transient haemoptysis associated with diagnostic bronchoscopy is allowed.
   3. Nasal bleeding /epistaxis (bloody nasal discharge is allowed).
   4. Need for therapeutic anticoagulant therapy within 14 days prior to randomization.

   Note: Prophylactic anticoagulation for deep vein thrombosis or pulmonary embolism or to maintain venous patency is allowed.
8. Current hypertension with systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg after oral antihypertensive therapy.
9. History of major diseases before randomization, specifically:

   1. Unstable angina, myocardial infarction, congestive heart failure (New York Heart Association classification ≥ grade 2) or vascular disease (eg, aortic aneurysm at risk of rupture) that required hospitalization within 12 months prior to randomization, or other cardiac impairment that may affect the safety evaluation of the study drug (eg, poorly controlled arrhythmias, myocardial ischemia),
   2. History of oesophageal gastric varices, severe ulcers, wounds that do not heal, abdominal fistula, intra-abdominal abscesses, or acute gastrointestinal bleeding within 6 months before randomisation,
   3. History of arterial thromboembolic event, venous thromboembolic event of Grade 3 and above as specified in NCI-CTCAE v5.0, transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy within 6 months prior to randomization,
   4. Acute exacerbation of chronic obstructive pulmonary disease within 4 weeks before randomisation,
   5. History of perforation of the gastrointestinal tract and/or fistula, history of gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection) within 6 months prior to randomisation.
10. Imaging during the screening period shows that the patient has:

    1. Radiologically documented evidence of major blood vessel invasion or encasement by cancer,
    2. Radiographic evidence of intra-tumour cavitation.
11. Microsatellite instability positive disease.
12. Concurrent malignancy (other than advanced biliary tract cancer), with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin. Cancer survivors, who have undergone potentially curative therapy for a prior malignancy, have no evidence of that disease for 5 years or more and are deemed at negligible risk for recurrence, are eligible for the trial.
13. HIV positive (HIV 1/2 antibodies patients), or a known history of active Tuberculosis bacillus.
14. Any immunosuppressive therapy (i.e. corticosteroids >10mg of hydrocortisone or equivalent dose) within 14 days before the planned start of study therapy.
15. Active autoimmune disease that has required a systemic treatment in past 2 years (i.e. corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin) is allowed active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

    1. Patients with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone are eligible for the study,
    2. Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study,
    3. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

       * Rash must cover < 10% of body surface area,
       * Disease is well controlled at baseline and requires only low-potency topical corticosteroids,
       * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months.
16. Prior allogeneic bone marrow transplantation or prior solid organ transplantation.
17. Any condition which in the Investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol.
18. Pregnant or breast-feeding females.
19. Participation in another therapeutic trial within the 30 days prior to entering the study. Participation in an observational trial would be acceptable.
20. Patients unwilling or unable to comply with the medical follow-up required by the trial because of geographic, familial, social, or psychological reasons.
21. Individuals deprived of liberty or placed under protective custody or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2027-08-03 (Estimated); Study Completion 2029-01-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From randomisation to disease progression or death, up to 4 years
  The progression-free survival is the length of time during and after the treatment of a disease that a patient lives with the disease but it does not get worse.

SECONDARY OUTCOMES:
Overall Survival (OS) | From randomisation to death, up to 4 years
  The overall survival is the length of time from randomization that patients enrolled in the study are still alive.
Objective response rate | From randomisation, up to 4 years
  The proportion of patients achieving complete response (CR) or partial response (PR) (according to RECIST v1.1). Objective response rate will be presented as the best response achieved compared to the disease assessment performed at randomisation.
Disease control rate | From randomisation, up to 4 years
  The proportion of randomised patients achieving CR, PR, stable disease (SD) as assessed by the investigator according to RECIST v1.1
Duration of response | From response to disease progression or death, up to 5 years
  The time from first documented response (compared to baseline measurement taken at randomisation) until the date of disease progression, as assessed by the investigator according to RECIST v1.1, or death from any cause whichever occurs first.

OTHER OUTCOMES:
Quality of life questionnaire - Core 30 (QLQ-C30) | From baseline, every 2 cycles (every 4-6 weeks) until end of treatment, an average of 1 year
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of life Questionnaire - Biliary tract cancer module (QLQ-BIL21) | From baseline, every 2 cycles (every 4-6 weeks) until end of treatment, an average of 1 year
  This EORTC cholangiocarcinoma and gallbladder cancer specific questionnaire is intended to supplement the QLQ-C30.
  The QLQ-BIL21 contains 21 items to assess symptoms. 3 single-item assessments relating to treatment side effects, difficulties with drainage bags/tubes and concerns regarding weight loss, and 18 items grouped into 5 scales: eating symptoms (4 items), jaundice symptoms (3 items), tiredness (3 items), pain symptoms (4 items) and anxiety symptoms (4 items). All items are rated on a four-point Likert-type scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), and are linearly transformed to a 0-100 scale, with higher scores indicating more severe symptoms.
Incidence of Adverse Events | From randomisation, up to 4 years
  Safety and tolerability of the treatment will be evaluated using the National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5). NCI-CTCAE is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Julien Edeline, MD, Principal Investigator — Centre Eugène Marquis; Ivan Borbath, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain; John Bridgewater, MD, Principal Investigator — University College London Cancer Institute; David Malka, MD, Principal Investigator — Institut Mutualiste Montsouris
Locations (3):
- France (2):
  - Institute Mutualiste Montsouris, Paris
  - Centre Eugène Marquis, Rennes
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Unicancer will share de-identified individual data that underlie the results reported. A decision concerning the sharing of other study documents, including protocol and statistical analysis plan will be examined upon request.
Supporting Information: Study Protocol, SAP
Time Frame: Unicancer will consider access to study data upon written detailed request sent to Unicancer, from 6 months until 5 years after publication of summary data.
Access Criteria: The data shared will be limit to that required for independent mandated verification of the published results, the applicant will need authorization from Unicancer for personal access, and data will only be transferred after signing of a data access agreement.